CLINICAL TRIAL: NCT05910931
Title: Prospective Study for the Evaluation of the Efficacy and Concordance of Angiography With Indocyanine Green in the Identification of Complications After Oncoplastic Surgery and Skin and Nipple-skin Sparing Mastectomy
Brief Title: Efficacy of Angiography With Indocyanine Green in the Identification of Complications After Breast Surgery
Status: Recruiting | Type: Observational
Sponsor: University Hospital A Coruña (Other)
Responsible Party: Principal Investigator, Benigno Acea, Breast Surgeon, University Hospital A Coruña
Other Study IDs: gBreast 22
Record Dates: First submitted 2023-06-04; First posted 2023-06-20 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Skin Necrosis; Complication
Keywords: breast cancer; oncoplastic surgery; breast reconstruction; skin sparing mastectomy; nipple-skin sparing mastectomy; indocyanine color green
MeSH Terms: conditions — Necrosis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing ICG angiography: All women operated on in the breast unit who require a reduction mammoplasty, a skin-sparing mastectomy (or skin and nipple) with immediate reconstruction and local flaps for remodeling or implant coverage.
  Interventions: Drug: ICG angiography

INTERVENTIONS:
Drug: ICG angiography — * A first injection with the patient asleep before starting the intervention to visualize the vascular anatomy of each patient and assess the pedicles and incisions.
  * A second bolus after breast resection to assess the viability of skin flaps and glandular pedicles.
  * A third injection to obtain an angiography after implant placement and wound closure.
  For angiography, the SPY System with the SPY-Q software will be used.

SUMMARY:
During the performance of oncoplastic surgery and skin-sparing or skin-nipple mastectomy there is a significant loss in the perfusion of the cutaneous envelope of the breast, which can produce areas of vascular suffering of the skin that sometimes cause necrosis of the same. Skin necrosis is the most important adverse event in oncoplastic and reconstructive surgery of the breast, since it causes delays in adjuvant treatments to surgery, worsening of the cosmetic result, and, on occasions, loss of the implant and reconstruction.

Indocyanine color green (ICG) angiography has been proposed as a diagnostic alternative to determine the vascular perfusion of the skin envelope of the breast during surgery, which would allow the removal of tissue at risk of necrosis to avoid this complication during the postoperative period. However, the scientific literature does not currently allow an adequate assessment of this diagnostic procedure due to the absence of prospective studies that have evaluated its sensitivity, specificity, and predictive values.

The objective of this prospective study is to evaluate ICG angiography of skin flaps of the breast and the surgeon's decision in women with breast cancer or at high risk for breast cancer undergoing oncoplastic surgery or mastectomy with the help of skin or skin-nipple. Based on the results of this study, the sensitivity, specificity, and predictive values of this technique for the prediction of adverse events during the postoperative period will be established.

DETAILED DESCRIPTION:
Currently, surgery is a decisive therapeutic element in the management of women with breast cancer and at high risk for breast/ovarian cancer. In the first scenario, oncological surgery has evolved towards more complex technical procedures, such as oncoplastic surgery or skin-nipple-sparing mastectomies. These procedures have improved the quality of breast conservation or breast reconstruction, but have also increased the incidence of postoperative complications. In the second scenario, risk reduction mastectomies also share this same problem with an increase in adverse events after the use of ultra-conservative mastectomies. Without a doubt, skin necrosis is the most significant adverse event during the postoperative period in these patients due to three reasons. The first focuses on patients with breast cancer in whom skin necrosis delays the start of adjuvant treatments to surgery, chemotherapy or radiotherapy, causing greater complexity in their care process. Secondly, a significant number of these women with skin necrosis will require a second surgery to close the defect in the skin coverage, generally using a local flap, increasing care saturation and healthcare costs. Finally, these skin necrosis generate anatomical defects that in many cases will lead to cosmetic sequelae, worsening satisfaction and quality of life in this group of women. These consequences are especially relevant in women with prepectoral breast reconstruction, since the absence of muscle between the skin and the implant facilitates the exposure of the latter and, on occasions, the loss of the reconstruction.

During the last 15 years our unit has published various articles analyzing adverse events during the postoperative period in patients with oncoplastic, reconstructive and risk reduction surgery. Thus, in a comparative study between lumpectomy and oncoplastic surgery in patients in our unit, an incidence of skin necrosis of 2.5% was demonstrated in oncoplastic procedures compared to 0.1% in lumpectomy. This higher incidence of complications had a significant impact on the delay for the start of radiotherapy, increasing this delay by 10 days compared to the group with lumpectomy. In the context of mastectomy, our unit has recently published the results of its prospective study PreQ 20 and it has shown an incidence of 5.6% of necrosis and skin dehiscence in women with skin-sparing mastectomy and breast cancer. Finally, another prospective study identified technical complexity and the appearance of postoperative complications as the two variables related to the appearance of cosmetic sequelae during follow-up in patients in our unit. These results highlight the value of prevention and/or early identification of skin ischemia to reduce the rate of necrosis during the postoperative period, guarantee delays during the care process, reduce cosmetic sequelae, and increase satisfaction and quality of life for women. with breast cancer and/or at high risk.

Various studies have evaluated ICG angiography as a diagnostic method in mastectomy skin flap perfusion. To our knowledge, only two nonrandomized prospective studies have evaluated the sensitivity, specificity, and predictive values of this technique. The study by Phillips et al evaluated this procedure in 51 immediate reconstructions with expanders for the prediction of postoperative skin necrosis. Sensitivity, specificity, positive (PPV) and negative (NPV) predictive value were 90%, 50%, 56% and 88%, respectively. On the other hand, in the study by Munabi et al these values were 88%, 83%, 44% and 98%, respectively. In this latter study the authors found that smoking and epinephrine injection decreased the specificity of this diagnostic method from 98% to 83%. These studies have two limitations. The first refers to the fact that they have been performed in patients with a retropectoral breast reconstruction and through the use of expanders. Currently this type of reconstruction has been replaced by prepectoral reconstruction with direct implantation and for this reason we lack information on this new surgical modality. On the other hand, there are no studies that have evaluated ICG angiography in women with oncoplastic procedures.

A Cochrane Library review was recently published whose objective was to evaluate the capacity of ICG angiography for the prevention of necrosis in mastectomy skin flaps in women undergoing immediate reconstruction after skin-sparing mastectomy. In this review we found nine studies that compared the number of postoperative complications in women undergoing ICG breast skin assessment versus clinical assessment. In these studies, a total of 1,589 women with 2,199 breast reconstructions were evaluated, and the number of complications per patient or per breast was reported. The main patient-related results of this review were that:

* ICG can reduce reoperation rates.
* there is uncertainty as to whether ICG decreases the rates of mammary skin necrosis, infection, hematoma and seroma.

The main results referring to the breast were:

* ICG can reduce mammary skin necrosis, reoperation rates and infection.
* there is uncertainty as to whether ICG has an effect on hematoma and seroma rates. The evidence from the studies evaluated during this review is considered to be of very low quality as there are no prospective randomized studies. This review emphasizes the need for prospective studies to further investigate the use of the ICG in oncoplastic and reconstructive surgery of the breast.

These uncertainties have encouraged us to carry out this prospective study in order to evaluate the role of indocyanine green angiography in the intraoperative identification of skin areas at risk for the appearance of necrosis in the skin cover of the breast in women operated on by an immediate oncoplastic or reconstructive procedure. Usually, when we talk about a diagnostic procedure such as ICG angiography, its sensitivity, specificity, positive predictive value, and negative predictive value are described. These parameters reflect the characteristics of the diagnostic test and serve to decide when they should be used (sensitivity and specificity of the test) or what is the meaning of this test in a particular patient. Unfortunately, the scientific literature has not evaluated these parameters for ICG angiography in the context of prepectoral reconstruction and oncoplastic surgery, which leads to empirical use of this procedure. The ultimate goal of this study is to provide information on the sensitivity, specificity, and predictive values of ICG angiography in these two clinical settings. With this, we intend to identify those patients in whom this diagnostic procedure provides added value in their surgical planning, reducing the incidence of skin necrosis and other associated surgical complications.

ELIGIBILITY:
Inclusion Criteria:

The study population includes two type of patients:

* Women who underwent oncoplastic procedures for breast conservation. This group is made up of women with breast cancer in whom the Breast Unit tumor committee recommended a breast-conserving surgical procedure. The techniques included for this study are vertical mammoplasty, horizontal mammoplasty, and local flaps by displacement or rotation.
* Women undergoing a skin or skin/nipple-sparing mastectomy with immediate breast reconstruction. This group is made up of patients with a diagnosis of breast carcinoma, who require a mastectomy as surgical treatment, as well as those high-risk women whose mastectomy is aimed at reducing the risk of breast cancer. The surgical techniques included in this group are Carlson type 1, 2, 3 and 4 skin-sparing mastectomies and nipple and skin-sparing mastectomies using inframammary and vertical approaches. In all patients, the type of breast reconstruction will be the placement of a definitive implant in the prepectoral position.

Exclusion Criteria:

- Women with iodine allergy or thyroid disease are excluded from this study.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women operated on for breast cancer or risk-reducing surgery who underwent oncoplastic surgery or skin-sparing mastectomy were included. The study aims to assess the sensitivity and specificity of indocyanine color green to predict skin necrosis
Sampling Method: Non-Probability Sample
Enrollment: 221 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, and predictive values intraoperatory. | during surgery
  To assess the sensitivity, specificity, and predictive values of VIC angiography for intraoperative detection of skin areas at high risk for necrosis.
Sensitivity, specificity, and predictive values for postoperative complications | up to 1 month
  To evaluate the sensitivity, specificity, and predictive values of VIC angiography for the prediction of complications during the postoperative period (infection, seroma, hematoma, implant exposure, implant loss, reoperation).

SECONDARY OUTCOMES:
Vascularity of nipple areola complex | before surgery
  To assess the presurgical ability of IVC angiography to identify dominant vascularity of the nipple-areola complex.
Surgical planning | before surgery
  To assess the impact of IVC angiography on changing incision planning or surgical pattern.
Time | during surgery
  Identify the time from injection to visualization on the SPY that best predicts necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Benigno Acea Nebril, MD PhD, Principal Investigator — University Hospital A Coruña
Locations (1):
- Hospital Abente y Lago, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No